CLINICAL TRIAL: NCT03166787
Title: Hookah Smoking, Carbon Monoxide, and Coronary Endothelial Function
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the Pandemic and the nature of this study we decided to terminate this study.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Florian Rader, Staff Physician I, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Protocol 47441; R21DA041596 (NIH)
Record Dates: First submitted 2017-03-30; First posted 2017-05-25 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Smoking; Endothelial Dysfunction
MeSH Terms: conditions — Smoking | interventions — Tobacco Products; Ascorbic Acid; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Myocardial Blood Flow (Experimental): Myocardial contrast echocardiography will be used to measure regional myocardial perfusion .
  Interventions: Other: Charcoal hookah; Other: E-coal hookah; Other: Cigarette
- Assess Coronary Endothelial Function (Experimental): young hookah smokers will be randomized to have coronary endothelial function assessed before and after inhaling Carbon Monoxide or room air from a Douglas bag.
  Interventions: Drug: Carbon Monoxide inhalation; Other: Room Air inhalation
- Test coronary endothelial function (Experimental): Test coronary endothelial function before after hookah smokers smoke charcoal-heated hookah and before and after age-matched cigarette smokers smoke 2 cigarettes. In the same subjects, we will test for acute smoking-induced changes in LV wall strain by speckle tracking. Finally, in a subset of subjects we will repeat the MCE and speckle tracking studies after pretreatment with either i.v. vitamin C or one dose of oral tadalafil.
  Interventions: Drug: vitamin C; Drug: tadalafil

INTERVENTIONS:
Other: Charcoal hookah — The Myocardial Blood Flow (MBF) will be measured at rest and during the last minute of a 3-minute bout of handgrip at 30% Maximal voluntary contraction. This sequence will be performed before and after 12 young hookah smokers are randomized to smoke the same popular Starbuzz tobacco product heated with either charcoal for 30 min each.
  Arms: Myocardial Blood Flow
Other: E-coal hookah — The Myocardial Blood Flow (MBF) will be measured at rest and during the last minute of a 3-minute bout of handgrip at 30% Maximal voluntary contraction. This sequence will be performed before and after 12 young hookah smokers are randomized to smoke the same popular Starbuzz tobacco product heated with electrically (Global First "e-coal," ) for 30 min each.
  Arms: Myocardial Blood Flow
Other: Cigarette — The Myocardial Blood Flow (MBF) will be measured at rest and during the last minute of a 3-minute bout of handgrip at 30% Maximal voluntary contraction. This sequence will be performed before and after 12 young cigarette smokers smoke 2 cigarettes down to the stub over 30 min (to simulate real-world use).
  Arms: Myocardial Blood Flow
Drug: Carbon Monoxide inhalation — A subset (n=8) of the young hookah smokers will return on a later day and will be randomized to have coronary endothelial function assessed before and after inhaling 0.3 CO gas from a Douglas bag.
  Arms: Assess Coronary Endothelial Function
Other: Room Air inhalation — A subset 8 of the young hookah smokers will return on a later day and will be randomized to have coronary endothelial function assessed before and after inhaling room air from a Douglas bag.
  Arms: Assess Coronary Endothelial Function
Drug: vitamin C — in a subset of 6 subjects the study team will repeat the Myocardial Contrast Echocardiography and speckle tracking studies after pretreatment with either i.v. vitamin C .
  Arms: Test coronary endothelial function
Drug: tadalafil — in a subset of 6 subjects the study team will repeat the Myocardial Contrast Echocardiography and speckle tracking studies after pretreatment with one dose of oral tadalafil.
  Arms: Test coronary endothelial function

SUMMARY:
Hookah (water pipe) smoking is a new global epidemic. The World Health Organization wants to prohibit all claims that hookah is less harmful than cigarettes and wants hookah products to bear the same warning labels as cigarettes. But there is little scientific evidence to substantiate this proposal. Cigarettes, cigars, medicinal nicotine, and e-cigarettes all acutely impair brachial artery endothelial function (flow-mediated dilation, FMD). Also, cigarettes cause both acute and chronic impairment in coronary endothelial function, but the comparative effects of hookah are unknown. Hookah tobacco is heated with burning charcoal. So, the smoke contains "tar" and nicotine plus charcoal combustion products. These include carbon monoxide (CO) and proatherogenic oxidants (especially carbon-rich nanoparticles) that the study team expected to impair endothelial function.

DETAILED DESCRIPTION:
Hookah (water pipe) smoking is a new global epidemic. The World Health Organization wants to prohibit all claims that hookah is less harmful than cigarettes and wants hookah products to bear the same warning labels as cigarettes. But there is little scientific evidence to substantiate this proposal. Cigarettes, cigars, medicinal nicotine, and e-cigarettes all acutely impair brachial artery endothelial function (flow-mediated dilation, FMD). Also, cigarettes cause both acute and chronic impairment in coronary endothelial function, but the comparative effects of hookah are unknown. Hookah tobacco is heated with burning charcoal. So, the smoke contains "tar" and nicotine plus charcoal combustion products. These include carbon monoxide (CO) and proatherogenic oxidants (especially carbon-rich nanoparticles) that the study team expected to impair endothelial function. Surprisingly, in young hookah smokers, the study team found that hookah smoking is a potent acute stimulus to augment-not impair-FMD. And the enhanced FMD is caused by one or more charcoal combustion products: when the study team replaced charcoal in the hookah with a supposedly healthier electronic heat source ("e-coal"), FMD became acutely impaired just as with cigarettes. But brachial artery FMD is a poor index of coronary endothelial function. With hookah, the CO boost (10-fold larger than cigarettes) decreases hemoglobin (Hb) O2-carrying capacity, which will decrease myocardial O2 delivery unless offset by increased myocardial blood flow (MBF). Accordingly, the study team now turn our attention to acute and chronic effects of hookah smoking on coronary endothelial function.

BACKGROUND/SIGNIFICANCE Carbon monoxide (CO) is an endogenously produced gas that play important physiological roles in the circulation. Traditionally considered a poisonous gas that causes tissue hypoxia, CO produced by vascular cells as a byproduct of heme catabolism, also functions to regulate blood flow by inhibiting vasomotor tone, smooth muscle cells proliferation, and platelet aggregation. These vascular effects are thought to be mediated by cyclic guanosine monophosphate (cGMP) because both clinical observations and experimental data provide precedent that CO, like nitric oxide, constitutes a cGMP-dependent vasodilator. Drugs that upregulate the endogenous production of CO by heme oxygenase, such as CO releasing molecules (CORMs), are being developed to treat several vascular diseases.

The toxicity of CO is dependent on the: (1) gas concentration; (2) duration of exposure; and (3) whether exposures are intermittent or continuous. After CO is inhaled by the lungs, it reaches the blood stream where it is bound by hemoglobin, forming carboxyhemoglobin. Thus, serum carboxyhemoglobin levels, as a percentage of total hemoglobin, is a determining factor that correlate with the degree of CO intoxication and severity of symptoms. Continuous CO inhalation is fatally toxic at concentrations of 800 parts per million (ppm) or 0.08% in the air. Based on environmental science literature (not controlled clinical research studies), death occurs from continuous CO inhalation for 2-3 hours as with gas-fired kitchen ranges. Studies conducted in controlled research setting have demonstrated that intermittent CO inhalation for 1 hour at low doses (<250 ppm) offers protection against inflammation and ischemic injury in the heart, liver, and kidney. According to a recent study published in Nature, repeated exposures of 250 ppm of CO for 1 hour inhibit experimental atherosclerosis by a cGMP-dependent process in rats. Other studies have also demonstrated that exogenous CO causes cGMP-dependent vasodilation in isolated vascular rings, and, in intact animals, can augment nitric oxide-dependent vasodilation.

Initial studies by our group allowed us to discover that, in young healthy hookah smokers, hookah smoking is a potent acute stimulus to augment-not impair-endothelial function measured by brachial artery flow mediated dilation (FMD). The data implicate a pivotal mechanistic role of one or more charcoal combustion products in the augmented endothelial function: when burning charcoal was replaced with a healthier electronic heat source ("e-coal"), FMD became acutely impaired just as with cigarettes and almost all other known tobacco products including electronic-cigarettes. Interestingly, the CO boost after our hookah subjects smoked charcoal-heated hookah tobacco was ~10-fold higher than after smoking a cigarette (25+11 vs. 3+2 ppm). Tobacco literature provide evidence that the repeated CO exposure from cigarette smoking is associated with a reduced risk of pre-eclampsia (associated with pathological vasoconstriction) in pregnant women as compared with both non-smokers or users of smokeless tobacco (snuff) which does not generate CO.

Recently published studies by our study consultants showed that intermittent 0.12-0.15% CO inhaled by healthy smokers, to achieve mean carboxyhemoglobin 5+1% (which is equivalent to exhaled CO levels of 30 ppm), had no significant effect on blood pressure, heart rate, plasma catecholamines, platelet aggregation or C-reactive protein, a marker of inflammation. Similarly, acute CO inhalation clinical research literature conducted in healthy subjects show that levels of 0.05-1.2% CO are safe and produced no symptoms, no adverse effects and no change in standard physiological measures such as blood pressure and heart rate (Table 1). The effects of low levels of CO on human endothelial function has yet to be determined.

ELIGIBILITY:
Inclusion Criteria:

* 21-25 y/o hookah smokers: smoked hookah > 12 times in the last 12 months.
* 21-25 y/o cigarette smokers: smoked >100 cigarettes and smoked in the last 30 days.
* 35-49 y/o hookah smokers: smoke hookah at least once per week for > 20 years.
* 35-49 y/o cigarette smokers: have > 20 pack-year cigarette smoking history.
* All subjects must have:

  * no history of illicit drug use or marijuana.
  * no evidence of cardiopulmonary disease by history or physical.
  * no diabetes with fasting blood glucose <100 mg/dl.
  * BP<140/90 mmHg.
  * resting heart rate<100 bpm.
  * BMI<30kg•m2.
  * no prescription medication.
  * normal EKG and echocardiogram.

Exclusion Criteria:

* suboptimal echocardiographic window.
* exhaled CO>10 ppm (smoking non-abstinence).
* positive pregnancy test.
* psychiatric illness.
* other conditions deemed unsafe to participate.

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
the change in Myocardial Blood Flow. | 90 minute
  the change in Myocardial Blood Flow between Baseline and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Victor, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No